CLINICAL TRIAL: NCT04410900
Title: Rabies Vaccination to Assess Vaccine Responsiveness After B Cell Targeted CAR-T Cell Therapies
Brief Title: Vaccine Responsiveness After CAR-T Cell Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG1007238; NCI-2020-03444 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10411 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: B-Cell Neoplasm
Keywords: CAR T cells; infection; vaccine; immunity
MeSH Terms: conditions — Lymphoma, B-Cell; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (anti-rabies vaccine, collection of blood) (Experimental): BOLUS COHORT: Patients receive the inactivated rabies vaccine IM on day 1 and 6-10 weeks later. Patients also undergo a blood collection prior to each vaccine, and at approximately 1, 2, and 4 weeks after each vaccination. A final blood collection occurs 6 months after the first immunization.
  FRACTIONAL DOSE COHORT: Patients receive the inactivated rabies vaccine fractionated primary dose IM on days 1, 3, 7, 10, 14, and 17 and the second dose 6-10 weeks later. Patients also undergo a blood collection prior to each vaccine, and at approximately 1, 2, and 4 weeks after each vaccination. A final blood collection occurs 6 months after the first immunization.
  Interventions: Biological: Wistar Rabies Virus Strain PM-1503-3M Vaccine; Procedure: Biospecimen Collection
- Control (anti-rabies vaccine, collection of blood) (Active Comparator): Patients receive anti-rabies vaccine IM on day 1 and 6-10 weeks later. Patients also undergo collection of blood samples at baseline, and at approximately 1, 2, and 4 weeks after each vaccination. There will be an additional blood draw 6 months (+/- 14 days) after the first immunization.
  Interventions: Biological: Wistar Rabies Virus Strain PM-1503-3M Vaccine; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Wistar Rabies Virus Strain PM-1503-3M Vaccine — Given IM
  Other Names: Imovax Rabies
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected

SUMMARY:
This phase I trial will use the inactivated rabies virus vaccine to assess immune function in patients who previously underwent B cell targeted chimeric antigen receptor-modified T cell immunotherapy (CARTx). A cohort of healthy volunteers will also be enrolled as a comparator group. CARTx is a new treatment for patients with B-cell malignancies (cancer of the B-cells), and the long-term effects of CARTx on immune function are not yet well understood. Learning more about vaccine responsiveness in patients who previously underwent CARTx may help doctors better understand immune function. The findings will guide evidence-based strategies for infection prevention to improve outcomes in this rapidly growing population of high-risk individuals.

DETAILED DESCRIPTION:
STUDY DESIGN:

This study will be a prospective, open-label clinical trial of primary and secondary vaccination with the inactivated rabies vaccine in patients treated with CARTx for B cell malignancies and healthy individuals. The target enrollment for this trial is 43 CARTx recipients and 10 healthy controls. The study is open to anyone regardless of gender or ethnicity.

OUTLINE:

BOLUS COHORT: Patients receive the inactivated rabies vaccine intramuscularly (IM) on day 1 and 6-10 weeks later. Patients also undergo a blood collection prior to each vaccine, and at approximately 1, 2, and 4 weeks after each vaccination. A final blood collection occurs 6 months after the first immunization. This will include up to 31 participants.

FRACTIONAL DOSE COHORT: Patients receive the inactivated rabies vaccine fractionated primary dose IM on days 1, 3, 7, 10, 14, and 17 and the second dose 6-10 weeks later. Patients also undergo a blood collection prior to each vaccine, and at approximately 1, 2, and 4 weeks after each vaccination. A final blood collection occurs 6 months after the first immunization. This will include up to 12 participants.

ELIGIBILITY:
Inclusion Criteria:

* CARTx RECIPIENTS: Patients must be capable of understanding and providing a written informed consent
* CARTx RECIPIENTS: Patients must be 18 years of age or older, of any gender, race or ethnicity
* CARTx RECIPIENTS: Patients must have had relapse-free survival for >= 6 months after receiving CARTx for B-cell malignancies
* CARTx RECIPIENTS: Platelet count > 30,000 / mm^3
* HEALTHY CONTROLS: Patients must be capable of understanding and providing a written informed consent
* HEALTHY CONTROLS: Patients must be 18 years of age or older, of any gender, race or ethnicity

Exclusion Criteria:

* CARTx RECIPIENTS: Patients who have received a hematopoietic cell transplant after CARTx
* CARTx RECIPIENTS: Previously received 1 or more rabies vaccines prior to the first vaccine visit
* CARTx RECIPIENTS: Patients who have received lymphodepleting therapies after CARTx and within the past 6 months
* CARTx RECIPIENTS: Patients with signs or symptoms of active infection
* CARTx RECIPIENTS: Patients who are pregnant or breastfeeding
* CARTx RECIPIENTS: Patients with previous known allergies to any component of the vaccine
* CARTx RECIPIENTS: Patients who have previously experienced a reaction to any vaccine that required medical attention
* CARTx RECIPIENTS: Study participants who report a severe adverse event following the first rabies vaccine will not be eligible for a second dose
* CARTx RECIPIENTS: Receiving corticosteroids > 0.5 mg/kg/day prednisone equivalence in the 7 days prior to first or second vaccination
* HEALTHY CONTROLS: Previously received 1 or more rabies vaccines
* HEALTHY CONTROLS: Chronic illness
* HEALTHY CONTROLS: Signs or symptoms of active infection
* HEALTHY CONTROLS: Pregnant or breastfeeding
* HEALTHY CONTROLS: Patients with previous known allergies to any component of the vaccine
* HEALTHY CONTROLS: Previous reaction to a vaccine that required medical attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with positive vaccine response | 4 weeks after the secondary vaccination
  This will be defined as a rabies virus neutralizing antibody (RVNA) titer ≥0.5 IU/ml at week 4 post-secondary immunization. This RVNA titer is considered to be evidence of an adequate immune response by the World Health Organization. Will estimate with 95% confidence intervals.

SECONDARY OUTCOMES:
Proportion of participants with sustained vaccine response | 6 months after the primary vaccination
  This will be defined as a rabies virus neutralizing antibody (RVNA) titer ≥0.5 IU/ml at 6 months following the primary vaccination in participants who also receive secondary vaccination per-protocol
Longitudinal rabies virus neutralizing antibody (RVNA) titers | From baseline (prior to primary vaccination) through 6 months after primary vaccination based on measurements at weeks 0, 1, 2, 4, 6, 7, 8, 10, and 24.
  Will compare quantitative levels of RVNA (log10 IU/mL) between CAR-T cell therapy and healthy participants at weekly intervals after each vaccination and at 6 months after primary vaccination.
Longitudinal rabies virus binding IgM antibody titers | From baseline (prior to primary vaccination) through 6 months after primary vaccination based on measurements at weeks 0, 1, 2, 4, 6, 7, 8, 10, and 24.
  Will compare quantitative levels of anti-rabies virus IgM between CAR-T cell therapy and healthy participants at weekly intervals after each vaccination and at 6 months after primary vaccination.
Longitudinal rabies virus binding IgG antibody titers | From baseline (prior to primary vaccination) through 6 months after primary vaccination based on measurements at weeks 0, 1, 2, 4, 6, 7, 8, 10, and 24.
  Will compare quantitative levels of anti-rabies virus IgG between CAR-T cell therapy and healthy participants at weekly intervals after each vaccination and at 6 months after primary vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A. Hill, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a future article will be shared, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared to achieve aims in the approved proposal. Proposals should be directed to Joshua A. Hill. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT04410900/ICF_000.pdf